CLINICAL TRIAL: NCT02339792
Title: Effect of an Integrated E-learning Intervention, Focused on Comprehensive Geriatric Assessment to Improve the Quality of Drug Prescribing in Hospitalized Elderly Patients
Brief Title: E-learning to Improve the Quality of Drug Prescribing in Hospitalized Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Paola Boccardo, MD, Mario Negri Institute for Pharmacological Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FARM87SA2B
Record Dates: First submitted 2014-12-16; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Drug Use
Keywords: COMPREHENSIVE GERIATRIC ASSESSMENT (CGA); MEDICATION APPROPRIATENESS PRESCRIBING; DRUG INTERACTIONS; E-LEARNING

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): e-learning program of medical education, focused on teaching and implementing Comprehensive Geriatric Assessment (CGA) added to geriatric pharmacological notions (GPNs)
  Interventions: Other: E-learning
- Control (Other): e-learning program of medical education, focused on teaching only geriatric pharmacological notions (GPNs)
  Interventions: Other: E-learning

INTERVENTIONS:
Other: E-learning — e-learning program of medical education, focused on teaching and implementing Comprehensive Geriatric Assessment (CGA) added to geriatric pharmacological notions (GPNs)

SUMMARY:
This randomized controlled pragmatic study is aimed to set-up, assess and implement an integrated e-learning program of medical education in an hospital setting, focused on teaching and implementing CGA added to geriatric pharmacological notions (GPNs) to improve the quality of drug prescribing in elderly patients

DETAILED DESCRIPTION:
The integrated e-learning program (intervention group) is focused on teaching and implementing knowledge on CGA and GPNs to help clinicians to improve the quality of drug prescribing in the elderly.The GPNs is focused on pharmaco-epidemiological issues of drug prescribing, pharmacokinetic and pharmacodynamic changes during aging, topics in evaluating and managing polypharmacy, criteria to review the appropriateness of drug therapies and the clinical relevance of PDDI in the elderly. The control group receives only GPNs.

ELIGIBILITY:
Inclusion Criteria:

* people aged 75 years or older

Exclusion Criteria:

* people aged 75 years or older
* refusal of consent to participate
* a life expectancy of less than 6 months

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 697 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Improvement of drug prescribing | Participants will be followed for the duration of hospital stay, an expected average of 12 days
  The primary study objective is to evaluate whether an integrated e-learning program of medical education, focused on teaching and implementing CGA added to GPNs (intervention) is superior to delivering GPNs only (control) in reducing the prescription of potentially inappropriate medications (PID) or of potential drug-drug interactions (PDDI) during hospitalization and at hospital discharge in hospitalized elderly.
  The primary outcome is the change in prescription of PID,as defined by Beers' criteria , or of PDDI related to the 20 drugs most frequently prescribed during hospital stay and at discharge.

SECONDARY OUTCOMES:
clinical outcomes (lenght of hospitalization, mortality, rehospitalization) | 12 months
  Secondary objectives are the assessment of:
  - the impact of the integrated e-learning intervention in terms of length of hospitalization, in-hospital and overall mortality, re-hospitalization and institutionalization during a follow-up of 12 months; - the persistence and the clinical impact on the enrolled patients of the effect of the integrated e-learning intervention on the improvement of quality of drug prescribing during a follow-up of 12 months.
  Secondary outcomes are the persistence and the clinical impact of the integrated e-learning intervention on duration of hospitalization, rate of in-hospital and overall mortality, re-hospitalization and institutionalization during 12 months of follow-up.

REFERENCES:
- [Derived] Franchi C, Tettamanti M, Djade CD, Pasina L, Mannucci PM, Onder G, Gussoni G, Manfellotto D, Bonassi S, Salerno F, Nobili A; ELICADHE Investigators. E-learning in order to improve drug prescription for hospitalized older patients: a cluster-randomized controlled study. Br J Clin Pharmacol. 2016 Jul;82(1):53-63. doi: 10.1111/bcp.12922. Epub 2016 Apr 5. PMID 26922904